CLINICAL TRIAL: NCT06750211
Title: Effects of Muscle Energy Techniques With and Without Motor Control Therapeutic Exercises on Pain, Range of Motion and Disability in Patients With Mechanical Neck Pain.
Brief Title: Effect of MET With and Without MCTE in Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0115
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Mechanical Neck Pain
Keywords: Neck pain; Range of motion; Muscle energy technique; Motor control therapeutic exercise
MeSH Terms: conditions — Neck Pain | interventions — ETV3 protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- METs (Active Comparator): Hot pack along with Neck isometrics and muscle energy technique protocol
  Interventions: Other: METs
- MCTE along with METs (Experimental): MCTE included cranio-cervical flexion, cranio-cervical extension, co-contraction of flexion and extension and synergistic exercise of neck flexor along with hot pack, neck isometrics and muscle energy technique protocol
  Interventions: Other: MCTE along with METs

INTERVENTIONS:
Other: METs — * Hot pack for 10 minutes.
  * Neck isometrics with 10 second hold.
  * Each series of neck isometrics strengthening exercises had three movements including cervical flexion, cervical extension and cervical side flexion.
  * Muscle energy technique protocol: The individual was in a position of supine. The therapist was at the edge of bed, near the participants head. the therapist positioned the joint at the point of beginning range of motion resistance when performing a given movement. When the therapist felt restriction, positioned the cervical spine in that region and apply the resistive force. Patient was instructed to contract isometrically for five seconds without exceeding the therapist force. thereafter, therapist counterforce gradually reduced and patient was asked to relaxed. Therapist move the joint into new point of barrier and same protocol repeated three times.
  Patient came thrice per week for a total of 4 weeks.
  Arms: METs
Other: MCTE along with METs — ▪ Hot pack for 10 minutes.
  * Neck isometrics with 10 second hold.
  * Each series of neck isometrics strengthening exercises had three movements including cervical flexion, cervical extension and cervical side flexion.
  * After it was treated with motor control therapeutic exercises together with muscle energy technique. Motor control therapeutic exercises included cranio-cervical flexor exercises, cranio-cervical extensor exercises, co contraction of flexor and extensor and synergy exercise for strengthening deep neck flexor. Exercises were performed in three sets with 10 repetitions with an approximate duration of 10 to 20 minutes. They were advised to perform at home once in a day, five times in a week for a duration of 4 weeks.
  All exercises were performed three times per week for total of 4 weeks.
  Arms: MCTE along with METs

SUMMARY:
Work had to be done previously on METs and MCTE techniques, but no study has compared both techniques together to make it more comprehensible. The rationale of this will be to find out the combined effect of motor control therapeutic exercises and muscle energy technique for the treatment of pain, range of motion and disability associated with mechanical neck pain. This study will be effective for the clinicians to treat patients of mechanical neck pain.

DETAILED DESCRIPTION:
Therapeutic exercises and manual therapy were shown to be useful in managing pain and lowering disability in patients with non-specific chronic neck pain (NCNP). However, little studies investigated the benefits of muscle energy technique and motor control therapeutics exercise on mechanical neck pain (MNP). The current research fulfill this gap by comparing the short and long term benefits of muscle energy technique with and without motor control therapeutic exercises (MCTE) with the grail of determining best approach for lowering pain and disability in mechanical neck pain patients.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects were between 20 and 50 years old.

  * Pain in cervical or neck region with no radiating pain in one or both upper limbs.
  * Pain minimum of 3 months.
  * Neck disability index (NDI) score of should be at least 10%.
  * Forward head posture.

Exclusion Criteria:

* • Neck pain associated with vertigo.

  * Irradiated neck pain.
  * Vertebral fracture.
  * Osteoporosis.
  * Previous neck injury.
  * Red flags (night pain, severe muscle loss, loss of involuntary control.
  * Subjects with difficulty in communication or understanding.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-08 (Estimated)

PRIMARY OUTCOMES:
Numeric pain scale rating | 4th week
  Changes from base line Pain intensity was assessed by Numeric Rating Scale (NRS). NRPS has fair to moderate reliability of test-retest in patients with Mechanical Neck Pain. The patient was required to indicate the number that represent his intensity of pain, in which 0 represents "no pain" and 10 represents "the worst pain imaginable". Numeric Pain Rating Scale is widely used subjective pain measure that has good test-retest reliability r = 0.79 - 0.96

SECONDARY OUTCOMES:
Neck disability index | 4th week
  Changes from base line NDI is self-assessment tool for the specific functional status of patients with neck pain, consisting of ten components pain, personal hygiene, obesity, reading, headache, focus, work, travelling, sleeping, and leisure, each part is scored on an index of 0 to 5, with 0 representing "painless" and 5 representing the "worst pain imaginable". These points earned are added to the total score. The questionnaire was determined in percentage. The NDI disability categories are: 0-8% without disability, 10-28% mild, 30-48% moderate, 50-64% serious, and 70-100% complete. NDI has fair to moderate reliability of test-retest in patients, with inter-class correlation coefficient ranging from 0.50-0.98.
ROM cervical spine (flexion) | 4th week
  Changes from base line Universal Goniometer is used for measuring neck range of motion. Reliability of goniometer was found for all the measurements ranging from, interclass correlation coefficient for goniometer > 0.94. The concurrent validity of goniometer was good with ICC value of > 0.85. The goniometer will be used to measure flexion.
ROM cervical spine (Extension) | 4th week
  Changes from base line Universal Goniometer is used for measuring neck range of motion. Reliability of goniometer was found for all the measurements ranging from, interclass correlation coefficient for goniometer > 0.94. The concurrent validity of goniometer was good with ICC value of > 0.85. The goniometer will be used to measure extension.
ROM cervical spine (Side flexion) | 4th week
  Changes from base line Universal Goniometer is used for measuring neck range of motion. Reliability of goniometer was found for all the measurements ranging from, interclass correlation coefficient for goniometer > 0.94. The concurrent validity of goniometer was good with ICC value of > 0.85. The goniometer will be used to measure side flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Rafique, phd, Principal Investigator — Riphah International University
Locations (1):
- Riphah college of rehabilitation and allied health sciences, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Letafatkar A, Rabiei P, Alamooti G, Bertozzi L, Farivar N, Afshari M. Effect of therapeutic exercise routine on pain, disability, posture, and health status in dentists with chronic neck pain: a randomized controlled trial. Int Arch Occup Environ Health. 2020 Apr;93(3):281-290. doi: 10.1007/s00420-019-01480-x. Epub 2019 Oct 25. PMID 31654125
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Martin-Gomez C, Sestelo-Diaz R, Carrillo-Sanjuan V, Navarro-Santana MJ, Bardon-Romero J, Plaza-Manzano G. Motor control using cranio-cervical flexion exercises versus other treatments for non-specific chronic neck pain: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2019 Jul;42:52-59. doi: 10.1016/j.msksp.2019.04.010. Epub 2019 Apr 20. PMID 31030111
- [Background] Parikh P, Santaguida P, Macdermid J, Gross A, Eshtiaghi A. Comparison of CPG's for the diagnosis, prognosis and management of non-specific neck pain: a systematic review. BMC Musculoskelet Disord. 2019 Feb 14;20(1):81. doi: 10.1186/s12891-019-2441-3. PMID 30764789
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164